CLINICAL TRIAL: NCT04275388
Title: Retrospective Cohort to Evaluate the Effectiveness and Safety of Xiyanping Injection Combined With Conventional Treatment for New Coronavirus Infection Pneumonia (Common Type)
Brief Title: Xiyanping Injection for the Treatment of New Coronavirus Infected Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: QF-XYP2001-1
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-04

CONDITIONS: 2019 Novel Coronavirus Pneumonia
MeSH Terms: interventions — Lopinavir; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — routine blood test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Xiyanping injection +other drugs: Drug: Xiyanping injection Xiyanping injection: 10-20ml daily, Qd, the maximum daily dose does not exceed 500mg (20mL) Other drugs: Lopinavir tablet or Ritonavir tablet;Alpha-interferon nebulization;Abidor Hydrochloride
  Interventions: Drug: Xiyanping injection; Drug: Lopinavir / ritonavir, alpha-interferon nebulization,Abidor Hydrochloride
- other drugs: Lopinavir tablet or Ritonavir tablet;Alpha-interferon nebulization;Abidor Hydrochloride
  Interventions: Drug: Lopinavir / ritonavir, alpha-interferon nebulization,Abidor Hydrochloride

INTERVENTIONS:
Drug: Xiyanping injection — Xiyanping injection, 10-20ml daily, Qd, the maximum daily does not exceed 500mg (20mL) + Lopinavir tablet /Ritonavir tablet or Alpha-interferon nebulization or Abidor Hydrochloride,
  Groups: Xiyanping injection +other drugs
Drug: Lopinavir / ritonavir, alpha-interferon nebulization,Abidor Hydrochloride — Lopinavir / ritonavir tablets, 2 times a day, 2 tablets at a time; alpha-interferon nebulization;Abidor Hydrochloride

SUMMARY:
the investigators conduct a randomized, open-label trial to evaluate and compare the safety and efficacy of Xiyanping injection in patients with 2019-nCoV pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory examination (RT-PCR) confirms the infection 2019-nCoV, which meets the diagnostic criteria for pneumonia (common type) in the New Coronavirus Infection Pneumonia Diagnosis and Treatment Program (Trial Version 6);
2. The patient has a complete hospitalization record that can be used for research.

Exclusion Criteria:

-

Subjects who meet any of the following criteria cannot be enrolled:

1. Suffering from diseases that need to be distinguished from pneumonia infected with new coronavirus, such as tuberculosis, bacterial or viral pneumonia other than new coronavirus pneumonia, hospital-acquired pneumonia, and other pathogenic microorganisms pneumonia;
2. People with basic diseases such as primary immunodeficiency disease, acquired immunodeficiency syndrome, congenital respiratory tract malformations, abnormal lung development, aspiration pneumonia, and lung malignant tumors;
3. According to the judgment of the investigator, the previous or current disease may affect the patient's participation in the trial or the outcome of the study, including: malignant disease, autoimmune disease, liver and kidney disease, blood disease, neurological disease, and endocrine Disease; presently suffering from diseases that seriously affect the immune system, such as: human immunodeficiency virus (HIV) infection, or blood system, or splenectomy, organ transplantation, etc;
4. Pneumonia diagnosed with severe, critically re-associated coronavirus infection or requiring mechanical ventilation or systemic anti-hormonal therapy;
5. Used Chinese patent medicines with similar efficacy as Xiyanping injection during the treatment.
6. The investigator judges that the relevant test or data is missing during the treatment process, which affects the research evaluation or analyst.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with new coronary pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 426 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-07-14 (Estimated); Study Completion 2021-12-14 (Estimated)

PRIMARY OUTCOMES:
Clinical recovery time | Up to Day 14
  From the beginning of study drug use to fever, respiratory rate, blood oxygen saturation to normal and cough relief, and maintained for at least 72 hours or more, calculated in hours

SECONDARY OUTCOMES:
Complete fever time | Up to Day 14
  From the beginning of research drug use to body temperature <37.3 ℃ (underarm) or mouth temperature ≤37.5 ° C, or anal or ear temperature ≤37.8 ° C, and maintained for 24h or more
Cough relief time | Up to Day 14
  Cough score "day + night" from the beginning of study medication to cough ≤ 1 point, and maintained for 24 hours and above
Virus negative time | Up to Day 14
  From the beginning of the study drug to two consecutive times (sampling interval of at least 1 day)
Incidence of severe or critical neocoronavirus pneumonia | Up to Day 14
  Defined as the proportion of subjects exacerbated during treatment and meeting the diagnostic criteria for severe or critical neocoronavirus pneumonia

IPD SHARING:
Plan to Share IPD: No